CLINICAL TRIAL: NCT02896660
Title: Activity Monitors for Opioid Dependence Treated With Probuphine
Brief Title: Probuphine Innovations for Clinical Effectiveness (PRINCE)
Acronym: PRINCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Healthcare Innovation Technology Lab (Industry)
Collaborators: Braeburn Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00018757
Record Dates: First submitted 2016-08-29; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-08

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ActiGraph Link (Experimental): Study participants will wear an actigraphy device, the ActiGraph Link, continuously for 90 days
  Interventions: Device: ActiGraph Link

INTERVENTIONS:
Device: ActiGraph Link — Subjects will be asked to wear the actigraph continuously for a 90-day period, and visit a clinician on day 30, 60, and 90 of the study for data collection.

SUMMARY:
HITLAB will conduct a crossover study wherein participants will be asked to wear an actigraphy device continuously for 12 weeks. The first four weeks of the study participants will continue their previously scheduled treatment regimen, prior to receiving the Probuphine implant. Following four weeks of activity and sleep baseline monitoring using the actigraphy device, the participant will receive the Probuphine implant as part of their regularly scheduled treatment plan. Observation of the participant's activity levels will continue for eight weeks following implantation of Probuphine. Actigraphy measurements will include total time asleep, total time awake, sleep efficiency, and time mobile.

DETAILED DESCRIPTION:
HITLAB will conduct a crossover study that measures the activity levels and sleep quality of patients both before and during treatment with Probuphine in order to determine whether Probuphine offers the additional benefit of improved energy levels during treatment, further distinguishing it from other opioid dependency treatments.

HITLAB researchers will meet with participating site physicians prior to study recruitment in order to administer the "Physician Baseline Questionnaire," a brief semi-structured baseline questionnaire to assess initial physician expectations for the actigraphy device.

Per physician guidelines, patients must be in stable treatment for at least 1 month prior to study enrollment. If the physician determines Probuphine to be an appropriate treatment method for the study subject, the physician will meet with the subject and explain the purpose of the actigraphy.

Upon enrollment, the physician will administer the "Participant Baseline Questionnaire," assessing general well-being, physical activity level, sleep patterns, and technology usage. At this time, the participant will be asked to begin wearing the Actigraph continuously for 12 weeks. The first four weeks of the study patients will continue their previously scheduled treatment regimen, prior to receiving the Probuphine implant.

Following four weeks of activity and sleep baseline monitoring using the actigraph device, the participant will receive the Probuphine implant [day 30]. At this visit, the clinician will administer four clinical assessments: Assessment of Withdrawal from Opioids Scale (SOWS), Clinical Opiate Withdraw Scale (COWS), Visual Analog Scales (VAS), and Measures of Morning Desire to use/need to use tool from Braeburn Pharmaceuticals (HS-11-421), as well as a baseline quality of life assessment (WHOQOL-BREF).

Observation of the participant's activity levels will continue for a total of eight weeks following implantation of Probuphine. Actigraphy measurements will include total time asleep, total time awake, sleep efficiency, and time mobile.

At the midline 60-day visit with each participant, as part of their regular monthly treatment appointment, the physician will repeat administration of the four clinical assessments (The Assessment of Withdrawal from Opioids Scale (SOWS), Clinical Opiate Withdraw Scale (COWS), Visual Analog Scales (VAS), and Measures of Morning Desire to use/Need to use tool from Braeburn Pharmaceuticals (HS-11-421)), as well as the quality of life assessment (WHOQOL-BREF).

At the participant endline visit [90 days], a physician will administer a repeat quality of life questionnaire (WHOQOL-BREF), and the four clinical assessments: Assessment of Withdrawal from Opioids Scale (SOWS), Clinical Opiate Withdraw Scale (COWS), Visual Analog Scales (VAS), and Measures of Morning Desire to use/need to use tool from Braeburn Pharmaceuticals (HS-11-421).

In addition, five participants will be randomly selected to participate in a short qualitative interview at the time of the site endline visit. Participant interviews, in person or via telephone, will assess their experience using the actigraph device during treatment, and their perspectives on activity changes and sleep quality. Patient perspectives on activity changes and sleep quality will serve as a point of triangulation for the actigraphy data.

HITLAB will conduct a baseline site visit, a site visit after 30 days, after 60 days, and after 90 days (the endline visit) of the study period to collect questionnaire and assessment data for analysis. Actigraphy data will be uploaded at days 30, 60 and 90. At the endline site visit, participating physicians will be asked to complete a brief, semi-structured "Physician Endline Questionnaire" to assess satisfaction with the actigraphy device in helping them improve outcomes and quality of life for patients in Probuphine treatment. A HITLAB researcher will also conduct a brief qualitative interview with the physicians at the endline site visit. The in-person physician interviews will assess whether the actigraphy data informed patient experience in such a way that it improves the efficacy of Probuphine administration and treatment.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must:

1. Be Adults over the age of 18
2. Speak English
3. In treatment for opioid addiction/dependence
4. Meet the criteria for treatment with Probuphine (on 8mg or less Subutex or Suboxone sublingual tablet or generic equivalent not requiring dose adjustment x 1 month)
5. Be clinically stable
6. Be willing to follow study procedures-including wearing a wearable actigraphy device-for 3 months

Exclusion Criteria:

Potential subjects must not:

1. Be less than 18 years of age
2. Do not meet the criteria for opioid dependence based on APA guidelines
3. Do not meet the criteria for treatment with Probuphine
4. Are not clinically stable or suffer from other mitigating issues surrounding addiction or psychological state.
5. Are not willing to follow study procedures-including wearing a wearable actigraphy device-for 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with changes in energy levels, as assessed by ActiGraph Link GT9X-BT | 90 days
  Patients will wear an actigraphy device to assess changes in activity over a 90-day period.

SECONDARY OUTCOMES:
Number of participants with changes in sleep quality, as assessed by ActiGraph Link GT9X-BT | 90 days
  Patients will wear an actigraphy device to assess changes in sleep quality over a 90-day period.
Number of participants with changes in quality of life, as assessed by WHOQOL-BREF | 90 days

OTHER OUTCOMES:
Number of participants with changes in self-reported desire/need to use symptoms, as assessed by Assessment of Withdrawal from Opioids Scale (SOWS) | 90 days
Number of participants with changes in clinician-reported desire/need to use symptoms, as assessed by Clinical Opiate Withdrawal Scale (COWS) | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Stan Kachnowski, PhD, Principal Investigator — Healthcare Innovation Technology Lab

IPD SHARING:
Plan to Share IPD: No
All participant data will be anonymous and reported in aggregate.

REFERENCES:
- [Background] Hartwell EE, Pfeifer JG, McCauley JL, Moran-Santa Maria M, Back SE. Sleep disturbances and pain among individuals with prescription opioid dependence. Addict Behav. 2014 Oct;39(10):1537-42. doi: 10.1016/j.addbeh.2014.05.025. Epub 2014 Jun 2. PMID 24999989
- [Background] Wilson KG, Watson ST, Currie SR. Daily diary and ambulatory activity monitoring of sleep in patients with insomnia associated with chronic musculoskeletal pain. Pain. 1998 Mar;75(1):75-84. doi: 10.1016/S0304-3959(97)00207-8. PMID 9539676
- [Background] Ancoli-Israel S, Cole R, Alessi C, Chambers M, Moorcroft W, Pollak CP. The role of actigraphy in the study of sleep and circadian rhythms. Sleep. 2003 May 1;26(3):342-92. doi: 10.1093/sleep/26.3.342. PMID 12749557
- [Background] Vallieres A, Morin CM. Actigraphy in the assessment of insomnia. Sleep. 2003 Nov 1;26(7):902-6. doi: 10.1093/sleep/26.7.902. PMID 14655927